CLINICAL TRIAL: NCT05750823
Title: An Open-Label, Phase 2, Safety, and Efficacy Study of Ruxolitinib Cream in Participants With Genital Vitiligo
Brief Title: A Study to Assess the Safety and Efficacy of Ruxolitinib Cream in Participants With Genital Vitiligo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB 18424-219; 2023-503737-22-00 (Registry Identifier: EU CT Number)
Expanded Access: NCT05722912 (Approved for marketing)
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Nonsegmental Vitiligo With Genital Involvement
Keywords: Vitiligo; Genital Vitiligo; INCB18424; Ruxolitinib Cream
MeSH Terms: conditions — Vitiligo | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib Cream (Experimental): Participants with non-segmental vitiligo with genital involvement will receive ruxolitinib 1.5% cream BID for up to 48 weeks
  Interventions: Drug: Ruxolitinib Cream

INTERVENTIONS:
Drug: Ruxolitinib Cream — Ruxolitinib cream will be applied twice daily for upto 48 weeks
  Other Names: Opzelura

SUMMARY:
An open-label study in which participants with non-segmental vitiligo with genital involvement will apply ruxolitinib 1.5% cream twice a day (BID) to all depigmented areas (up to 10% BSA) for up to 48 weeks. Participants should continue to treat depigmented areas identified for treatment at baseline regardless of whether the area begins to improve or fully repigment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of nonsegmental vitiligo with genital involvement
* At least ≥ 0.25% BSA of nonsegmental vitiligo in the genital area.
* Pigmented hair within some of the genital vitiligo areas.
* At least 1 genital target lesion that is ≥ 0.1% BSA that has a pigmented hair within it.
* Vitiligo on areas of the body besides the genitals.
* Total body vitiligo area not exceeding 10% BSA.
* Willing to have genital photography conducted.
* Must agree to discontinue all agents used to treat vitiligo from screening through the final safety follow-up visit. Over-the-counter preparations deemed acceptable by the investigator and camouflage makeups are permitted.

Exclusion Criteria:

* Other forms of vitiligo (eg, segmental) or other differential diagnosis of vitiligo or other skin depigmentation disorders.
* Prior or current use of depigmentation treatments (eg, monobenzone).
* Active or recurrent genital warts or herpes.
* Male participants with partners with known current/active cervical intraepithelial neoplasia or anal intraepithelial neoplasia.
* An active sexually transmitted disease, sexually transmitted infection, or other skin disorder affecting the genital area (eg, scabies, fungal infection, molluscum).
* Had ≥ 3 laser hair removal treatments in an area to be treated for vitiligo.
* Any serious illness or medical, physical, or psychiatric condition(s) that, in the investigator's opinion, would interfere with full participation in the study or interpretation of study data.
* Clinical laboratory test results outside of protocol defined ranges
* Pregnant or lactating participants, or those considering pregnancy during the period of their study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving a genital Vitiligo Noticeable Score (VNS) of 4 or 5 | Week 48
  Vitiligo Noticeable Score (VNS) is a patient-reported outcome measure on a scale of 1-5, 1- more noticeable, 4 - a lot less noticeable, and 5- no longer noticeable

SECONDARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | 52 weeks
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment.
Proportion of participants achieving Genital- Physician Global Vitiligo Assessment (PhGVA) | Week 48
  The severity of total body vitiligo will be assessed by the physician using the PhGVA on a scale of 0-4, 0 being clear to 4 being severe disease
Change from baseline in affected Body Surface Area BSA in the genital region | Week 24 and 48
  The BSA depigmented by vitiligo will be estimated at each visit.
Proportion of participants achieving T-VASI50/75/90 | Week 24 and 48
  ≥ 50%/75%/90% improvement in total body Vitiligo Area Scoring Index
Proportion of participants achieving a genital Vitiligo Noticeable Score (VNS) of 4 or 5 | Week 24
  Vitiligo Noticeable Score (VNS) is a patient-reported outcome measure on a scale of 1-5, 1- more noticeable, 4 - a lot less noticeable, and 5- no longer noticeable
Proportion of participants in each category of the color-matching question | Week 24 and 48
  Participants will answer how well the color of the treated skin matches the normal skin on a scale of 1-5, 1 being excellent to 5 being very poor.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (6):
  - Center For Dermatology Clinical Research, Inc, Fremont, California
  - Vitiligo & Pigmentation Institute of Southern California, Los Angeles, California
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Apex Clinical Research Center, Mayfield, Ohio
  - Austin Institute For Clinical Research Aicr Pflugerville, Pflugerville, Texas
  - Innovative Dermatology: Legacy Medical Village, Plano, Texas
- Canada (4):
  - Dermatology Research Institute, Calgary, Alberta
  - Simcomed Health Ltd, Barrie, Ontario
  - Skin Centre For Dermatology, Peterborough, Ontario
  - Research Toronto, Toronto, Ontario
- France (3):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Hopital Henri Mondor Service de Dermatologie, Créteil
  - Chu Nice Hopital Archet 2, Nice

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency